CLINICAL TRIAL: NCT00762138
Title: The AutoloGel™ Post-Market Surveillance (TAPS) Program
Acronym: TAPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinued due to favorable results
Sponsor: Cytomedix (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CM 306
Record Dates: First submitted 2008-09-24; First posted 2008-09-30 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Wounds; Leg Ulcers; Pressure Ulcers; Diabetic Foot Ulcers
Keywords: Platelet rich plasma; wounds; leg ulcers; pressure ulcers; diabetic ulcers; management of mechanically or surgically-debrided wounds
MeSH Terms: conditions — Wounds and Injuries; Leg Ulcer; Pressure Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologel System (Other): Autologel System produces platelet rich plasma gel
  Interventions: Device: AutoloGel System

INTERVENTIONS:
Device: AutoloGel System — The AutoloGel™ System may be used for chronic or surgically-debrided wounds up to twice a week for eight (8) weeks. The treating health care practitioner may elect to continue the treatment up to twelve (12) weeks. The AutoloGel™ System should be used in conjunction with standard of care procedures for comprehensive wound management , such as:
  Removal of necrotic or infected tissue Off-loading Compression therapy for venous stasis ulcers Establishment of adequate blood circulation Maintenance of a moist wound environment Management of wound infection Wound cleansing Nutritional support, including blood glucose control for subjects with diabetic ulcers Bowel and bladder care for subjects with pressure ulcers at risk for contamination Management of underlying disease
  Other Names: platelet-rich plasma (PRP) gel; such as leg ulcers, pressure ulcers, diabetic ulcers

SUMMARY:
AutoloGel™ Post-Market Surveillance Program

Purpose:Evaluate the incidence of hematologic and immunologic adverse events, including coagulopathies in patients with wounds to which AutoloGel™ was applied.

Design:Prospective, open label, patient registry. Investigator Sites: 3 Enrollment Size: 300

Subject Population: Patients with exuding wounds, such as leg ulcers, pressure ulcers, and diabetic ulcers and for the management of mechanically or surgically-debrided wounds.

Primary Objective Safety: Assess the incidence of hematologic (coagulopathies), immunologic (including anaphylaxis) and other adverse events associated with the application of AutoloGel on exuding wounds, such as leg ulcers, pressure ulcers and diabetic ulcers and during the management of mechanically or surgically-debrided wounds.

Primary Safety Endpoint: Absence of coagulopathies caused by inhibitors to coagulation Factor V as determined by a significant prolongation of the prothrombin (PT) time and confirmed by severe depletion of Factor V activity with a positive Bethesda Assay for anti-Factor V functional inhibitors.

DETAILED DESCRIPTION:
Device Name.

The device subject to the Post-Market Surveillance (PMS) Program is the AutoloGel™ System which has been cleared for marketing by the Food and Drug Administration (FDA) in the application BK060007.

The AutoloGel™ System includes.

AutoloGel™ Centrifuge II AutoloGel™ System Wound Dressing and Reagent Kits including single-use, disposable components for performing a patient phlebotomy, centrifuging blood to derive PRP and activating and applying the AutoloGel.

The Instructions for Use include a detailed description and procedures for making AutoloGel and a list of the Kit components which is provided at the end of the Instructions.

Indications for Use.

The AutoloGel™ System is intended to be used at point-of-care for the safe and rapid preparation of platelet-rich plasma (PRP) gel from a small sample of a patient's own blood. Under the supervision of a healthcare professional, the PRP gel produced by the AutoloGel™ System is suitable for exuding wounds, such as leg ulcers, pressure ulcers, and diabetic ulcers and for the management of mechanically or surgically-debrided wounds.

Dosing.

The AutoloGel™ System may be used for chronic or surgically-debrided wounds up to twice a week for eight (8) weeks. The treating health care practitioner may elect to continue the treatment up to twelve (12) weeks. The AutoloGel™ System should be used in conjunction with standard of care procedures for comprehensive wound management.

Removal of necrotic or infected tissue Off-loading Compression therapy for venous stasis ulcers Establishment of adequate blood circulation Maintenance of a moist wound environment Management of wound infection Wound cleansing Nutritional support, including blood glucose control for subjects with diabetic ulcers Bowel and bladder care for subjects with pressure ulcers at risk for contamination Management of underlying disease

Precautions and Warnings.

Caution. Federal Law (U.S.A.) restricts this device to sale by or on the order of a Physician.

Precautions.

Throughout the processing procedure and application of AutoloGel™, use universal precautions as defined by the facility policy and procedure manual.

All parts of the procedure shall be performed in such a manner to minimize splashing, spraying, spattering, and generation of potential droplets.

Warnings.

AutoloGelTM is produced with the use of bovine thrombin. The use of topical bovine thrombin preparations has occasionally been associated with abnormalities of hemostasis ranging from asymptomatic alterations in laboratory determinations, such as prothrombin time (PT) and partial thromboplastin time (PTT), to severe bleeding or thrombosis which have rarely been fatal. These hemostatic effects appear to be related to the formation of antibodies against bovine thrombin and / or factor V which in some cases may cross react with human factor V, potentially resulting in factor V deficiency. Repeated clinical applications of topical bovine thrombin increase the likelihood that antibodies against thrombin and / or factor V may be formed. Consultation with an expert in coagulation disorders is recommended if a patient exhibits abnormal coagulation laboratory values, abnormal bleeding or abnormal thrombosis following the use of topical thrombin. Any interventions should consider the immunologic basis of this condition. Patients with antibodies to bovine thrombin preparations should not be re-exposed to these products.

Allergic reactions may be encountered in persons known to be sensitive to bovine materials. Because of thrombin's action in the clotting mechanism, AutoloGel must not be injected or otherwise allowed to enter large blood vessels. Extensive intravascular clotting and even death may result.

ELIGIBILITY:
Inclusion Criteria:

* A patient who meets all the following criteria will be enrolled in the postmarket surveillance program:
* Presents with exuding wounds, such as leg ulcers, pressure ulcers, and diabetic ulcers and mechanically or surgically-debrided wounds.
* Male or female subject of any race, and 18 to 95 years old.

Exclusion Criteria:

* Study investigator(s) shall follow the Contraindications, Precautions, and Warnings relevant to subjects enrolled for treatment of wounds;
* Subjects will be excluded from the trial if any of the following criteria are met:
* If the Subject is on Coumadin medication (or another medication that is known to affect a potential coagulopathy) and has an elevated PT (prothrombin time) at the alert level at baseline, he/she will NOT be enrolled in the surveillance program.
* Ensure the patient does not have any Contraindications as noted in the AutoloGel System Instructions for use, specifically:
* Patients known to be sensitive to components and / or materials of bovine origin
* Patients on chemotherapeutic agents
* Patients with the following abnormal laboratory test levels

  * hemoglobin <10.5 g/dL
  * platelet count <100 x 109/L
  * serum albumin level < 2.5 g/dL
* Wounds due to malignancy
* Wounds with active clinically diagnosed infection

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Assess the incidence of hematological immunologic other ae's association with the application of AutoloGel on exuding wounds such as leg ulcers pressure ulcers and diabetics ulcers and during the management of mechanically or surgically debrided wounds | 3 years

SECONDARY OUTCOMES:
Absence of coagulopathies caused by inhibitors to coagulation Factor V as determined by a significant prolongation of the (PT) time. Depletion of Factor V activity with a positive Bethesda Assay | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Macy G Hall, MD, Principal Investigator — Speciality Hospital of Washington - Hadley; John G Martinez, MD, Principal Investigator — VA Southern Nevda; Janaki Nadarajah, DPM, Principal Investigator — Aiyan Diabetes Center; Gregory H Szeyko, MD, Principal Investigator — Providence Wound Institute
Locations (2):
- United States (2):
  - Aiyan Diabetes Center, Augusta, Georgia
  - Providence Wound Institute, El Paso, Texas

REFERENCES:
- See also: Related Info — http://www.cytomedix.com